CLINICAL TRIAL: NCT02519387
Title: Multicentre Study for Evaluation of the Efficacy and Safety of Buprenorphine Transdermal Patch (SOVENOR®) 5mg and 10mg in Patients With Non-malignant Pain of Moderate Intensity Due to Osteoarthritis, Rheumatoid Arthritis, Lower Back Pain and Joint/Muscle Pain, When an Opioid is Necessary for Obtaining Adequate Analgesia
Brief Title: Efficacy and Safety of Buprenorphine Transdermal Patch in Non-cancer Pain of Moderate Intensity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma Pharmaceuticals Sdn. Bhd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUP11-MY-401
Record Dates: First submitted 2015-07-15; First posted 2015-08-10 (Estimated); Results first posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Lower Back Pain; Joint Pain; Muscle Pain
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Low Back Pain; Arthralgia; Myalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Buprenorphine Transdermal Patch (Experimental): Buprenorphrine transdermal patch 5mg/10mg, every 7 days, for 3 months
  Interventions: Drug: Buprenorphine Transdermal Patch

INTERVENTIONS:
Drug: Buprenorphine Transdermal Patch
  Other Names: Sovenor®

SUMMARY:
This is a phase IV, open-label and single-arm study of patients with non-malignant pain due to osteoarthritis, rheumatoid arthritis, low back pain and joint/muscle pain, who were not responding to non-opioid analgesics. The primary objective was to assess the efficacy of buprenorphine transdermal patch for pain control among these patients.

DETAILED DESCRIPTION:
Buprenorphine transdermal (BTDs) is a semi-synthetic opioid analgesic. Earlier studies have shown BTDs to be non-inferior to an oral codeine-paracetamol combination and prolonged-release tramadol, in terms of pain control as well as sleep quality. BTDs is registered for use in Malaysia but the scientific data on efficacy and tolerability among Malaysians was not available. Thus, this study was conducted to evaluate the efficacy and tolerability of BTDs among Malaysian patients.

Patients eligible for entry into the study were adults aged ≥ 40 years who met the inclusion criteria and qualified from baseline screening and liver function test (LFT) assessment. The study excluded patients who met the exclusion criteria and failed prior the LFT assessment. Patients received an initial dose of 5 mg BTDs after qualifying on the baseline screening and LFT test. The dose could be up-titrated to a maximum of BTDs 20mg (2 X 10 mg) to achieve stable pain control.

There were six visits during the three-month study period. At visit 1, patients received 5mg of Sovenor® as initial treatment dose. Visit 2 occurred 7 days after the first visit; visit 2 and visit 3 were dose titration visits. Visit 4 and visit 5, were for assessment purposes. Primary treatment efficacy was measured during each visit with additional assessments of patients' sleep quality and quality of life, while physicians' and patients' treatment satisfaction assessed during the final visit. Safety was measured by monitoring the occurrence of adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 40 years and above at the time of recruitment.
2. Clinical diagnosis of osteoarthritis, rheumatoid arthritis, lower back pain or joint/muscle pain.
3. Having non-malignant pain of moderate intensity requiring an opioid for adequate analgesia. This was determined using BS-11 scores, where the cut-off point is ≥4.
4. Patients had to be opioid treatment naïve as defined by no opioid treatment (including tramadol, morphine etc.) in the preceding 1 month.
5. Patients who have uncontrolled pain and had not responded to non-opioid analgesics for 1 month or more.
6. Patients who provided informed consent.

Exclusion Criteria:

1. Pregnant and lactating females.
2. Patients with chronic condition(s), in addition to (osteoarthritis) OA, that required frequent analgesic treatment (e.g. frequent headaches, frequent migraine, and gout).
3. Patients who were awaiting a scheduled operation or other surgical procedure during study period.
4. Prior history of being on opioids in the preceding one month prior to the study for the management of chronic non-malignant pain.
5. Patients with history of allergic reactions against paracetamol/acetaminophen, Non Steroidal Anti-Inflammatory drugs (NSAIDs) and/or opioids.
6. Patients with allergies or other contraindications to transdermal systems or patch adhesives.
7. Patients with dermatological disorders who may have problems applying patch or rotating patch placement area.
8. Patients with cancer (except for basal cell carcinoma) or history of cancer who have been diagnosed within five years prior to the visit (except for treated basal cell carcinoma).
9. Patients with conditions such as brain tumour, brain injury or raised intracranial pressure.
10. Patients with history of psychiatric disorder, uncontrollable epilepsy, untreated depression or other psychiatric disorders of a type that would make participation in the study an unacceptable risk to the patient.
11. Patients with any conditions causing poor cognitive function as assessed by the participating physician.
12. Patients with history of alcohol and drug abuse or patients who had demonstrated behaviour that suggests a dependency or drug abuse.
13. Patients who were at the time taking hypnotics or other central nervous system depressants that may pose a risk of additional central nervous system (CNS) depression with study medication.
14. Patients who were at the time being administered monoamine oxidase inhibitors (MAOIs) or have taken MAOIs within 2 weeks before screening.
15. Patients who were at the time taking adjuvant analgesics such as anti-depressants (e.g. amitriptyline, amoxapine, clomipramine, selective serotonin re-uptake inhibitors (SSRIs)) and anticonvulsants (e.g. gabapentin, pregabalin).
16. Patients who had received steroid treatment (intra-articular, intramuscular, oral, intravenous, epidural or other corticosteroid injections) within 6 weeks prior to clinical study or planned steroid treatment during the clinical study period.
17. Patients who had to use heating facility over area of patch (examples: heating lamp, electric blanket, sauna, warm compresses, heated saline baths, etc.).
18. Patients who could not or did not wish to remove hair growing at body surface where the patch can be placed.
19. Any other contraindication mentioned in the Summary of Product Characteristics for Sovenor® transdermal patch.
20. Patients who were at the time on disability claims or in the process of applying for disability claims.
21. Patients at child-bearing age who were planning to conceive a child during the study period and were not practicing adequate contraception.
22. Patients with known severe hepatic impairment as determined by liver function test within the past one year. If liver function testing was not performed within 1 year prior to study initiation, patient had to undergo liver function testing prior to recruitment.
23. Patients who were at the time in or had participated in other clinical trials within the last 30 days prior to study recruitment.
24. Patients who were unable to comply to study visits.
25. Patients who, in the investigator's opinion, were not suited to participate in the study involving the study medicine for any other reason not stated in the inclusion/exclusion criteria.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Malaysia (3):
  - Hospital University Sains Malaysia, Kota Bharu, Kelantan
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - University Kebangsaan Malaysia Medical Centre, Kuala Lumpur, Kuala Lumpur

RESULTS

PARTICIPANT FLOW:
Groups:
- Buprenorphine Transdermal Patch: Buprenorphrine transdermal patch 5mg/10mg, every 7 days, for 3 months
  Buprenorphine Transdermal Patch
Period: Overall Study
Arm/Group | Buprenorphine Transdermal Patch
Started | 78
Completed | 56
Not Completed | 22

BASELINE CHARACTERISTICS:
Arm/Group | Buprenorphine Transdermal Patch
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 22
Region of Enrollment [Number; unit: participants]
  Malaysia | 78

OUTCOME MEASURES:

1. Primary Outcome: Change in Box Scale-11 (BS-11) Pain Score
Description: The BS-11 (Box score-11) pain score was the main efficacy outcome measured in this study. The scores at baseline (Visit 1) and Visit 6 (3 months from baseline visit) are reported.
  BS-11 is an 11-point scale measuring pain intensity. It ranges from 0 to 10, whereby 0 represents no pain and 10 represents the worst imaginable pain. Subjects selected a number based on the pain intensity they were feeling at that time.
Time Frame: Baseline,3 months
Population: These patients were eligible and included in the intent-to-treat efficacy population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine Transdermal Patch
Number analyzed (Participants) | 78
units on a scale
  Baseline (Visit 1) | 6.2 (1.8)
  3 Months (Visit 6) | 4.0 (2.3)

2. Secondary Outcome: Change in Sleep Quality as Determined by the 8-item Global Sleep Quality Assessment (GSQA)
Description: Subjects will evaluate the degree of their sleep disturbance due to pain and improvement in quality of sleep using the GSQA questionnaire comprising of 8 questions, at baseline (Visit 1) and Visit 6 (3 months from baseline visit).
  The scores at baseline and Visit 6 are calculated for the following 8 items with scores of:
  1. Trouble falling asleep due to pain -- on a scale of 0 to 10 where 0 is never and 10 is always
  2. Need for pain medication to sleep -- as above
  3. Need for sleep medication to sleep -- as above
  4. Awakened by pain at night -- as above
  5. Awakened by pain in the morning -- as above
  6. Pain affecting partner's sleep -- as above
  7. Rate own sleep quality -- on a scale of 1 to 5 where 1 is very good and 5 is very poor
  8. Number of hours of sleep per night in last 7 days
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine Transdermal Patch
Number analyzed (Participants) | 78
units on a scale
  Trouble falling asleep due to pain (Baseline) | 3.4 (2.9)
  Trouble falling asleep due to pain (3 Months) | 2.5 (2.9)
  Need for pain medication to sleep (Baseline) | 2.2 (2.9)
  Need for pain medication to sleep (3 Months) | 1.4 (2.5)
  Need for sleep medication to sleep (Baseline) | 0.3 (1.4)
  Need for sleep medication to sleep (3 Months) | 0.2 (1.2)
  Awakened by pain at night (Baseline) | 2.6 (2.8)
  Awakened by pain at night (3 Months) | 2.0 (2.6)
  Awakened by pain in the morning (Baseline) | 1.9 (2.5)
  Awakened by pain in the morning (3 Months) | 1.3 (2.3)
  Pain affecting partner's sleep (Baseline) | 1.2 (2.1)
  Pain affecting partner's sleep (3 Months) | 1.0 (2.0)
  Rate own sleep quality (Baseline) | 2.8 (0.8)
  Rate own sleep quality (3 Months) | 2.5 (0.8)
  Average hours of sleep per night (Baseline) | 5.7 (1.4)
  Average hours of sleep per night (3 Months) | 5.8 (1.4)

3. Secondary Outcome: Daily Use of Breakthrough Pain Medication as Measured by Number of Subjects With at Least 1 Day of Breakthrough (Rescue) Pain Medication Usage
Description: Patients will record any other pain medication used in a patient home diary
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Buprenorphine Transdermal Patch
Number analyzed (Participants) | 78
participants | 46

4. Secondary Outcome: Physicians' and Patients' Treatment Satisfaction of Buprenorphine Patch Usage Assessed Using Physician's Global Impression of Change Scale and Patient's Global Impression of Change Scale Respectively
Description: The overall assessment of the change in pain intensity from baseline is measured at Visit 6.
  Physician's Global Impression of Change scale: Investigator's opinion on a scale of 1 to 7 where 1 is "very much improved" and 7 is "very much worse" Patient's Global Impression of Change scale: Subject's opinion on a scale of 1 to 7 where 1 is "very much improved" and 7 is "very much worse"
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine Transdermal Patch
Number analyzed (Participants) | 78
units on a scale
  Physician Impression | 2.0 (0.7)
  Patient Impression | 2.3 (0.7)

5. Secondary Outcome: Tolerability of Buprenorphine Patch Determined by Number of Patients Who Withdrew From the Study Due to Adverse Events
Time Frame: 3 months
Population: This is the intent-to-treat population.
Measure: Number; unit: participants
Arm/Group | Buprenorphine Transdermal Patch
Number analyzed (Participants) | 78
participants | 17

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of 3 months from the time a patient is enrolled.
Arm/Group | Buprenorphine Transdermal Patch
Serious Adverse Events (participants affected / at risk) | 1/78
Other Adverse Events (participants affected / at risk) | 56/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine Transdermal Patch (N=78)
Elbow fracture due to fall (Musculoskeletal and connective tissue disorders) | 1 (1) — Hospitalisation
Failed elbow implant (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Buprenorphine Transdermal Patch (N=78)
Palpitation (Cardiac disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 14
Diarrhea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 22
Vomiting (Gastrointestinal disorders) | 10
Dry throat (Gastrointestinal disorders) | 2
Discomfort (General disorders) | 1
Drug intolerance (General disorders) | 1
Fatigue (General disorders) | 2
Myalgia (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 4
Peripheral swelling (General disorders) | 1
Application site allergy (Immune system disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 3
Hypoesthesia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 19
Somnolence (Nervous system disorders) | 17
Confusional state (Psychiatric disorders) | 1
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 15
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Increased blood pressure (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data emerging from the study cannot be released by the PI without permission from the sponsor.